CLINICAL TRIAL: NCT06255184
Title: Effect of Serenity Therapy on Symptoms Distress, Coping Styles, and Emotional Regulation Among Geriatric Patients Undergoing Hemodialysis: a Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mahmoud Khedr, Lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 93/2024
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Geriatric Patients

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serenity GROUP (Experimental): 40 geriatric patients for the serenity group. They will receive the routine care in addition to the serenity therapy which included 8 sessions (1 introductory session, 4 face to face sessions at dialysis unit , and 3 mobile based sessions at home).
  Interventions: Behavioral: Sernity intervention
- Control group (No Intervention): The control group received only the routine care provided at the dialysis unit with no extra interventions.

INTERVENTIONS:
Behavioral: Sernity intervention — Serenity Therapy is a holistic intervention that boosts psychological well-being and emotional balance through relaxation techniques, mindfulness, and guided imagery
  Arms: Serenity GROUP

SUMMARY:
Our research aims to examine the effect of the serenity therapy on symptoms distress, coping styles, and emotional regulation among geriatric patients undergoing hemodialysis. This study highlights the following question: what is the effect of the serenity therapy on symptoms distress, coping styles, and emotional regulation among geriatric patients undergoing hemodialysis.

DETAILED DESCRIPTION:
In order to conduct this study, a randomized controlled trial research design was followed. The selected sitting for this study was the hemodialysis unit of the National Medical Institute at Damanhur city, El-Behaira Governorate, Egypt. Geriatric patients who were recruited for this study, meet the following inclusion criteria; being sixty years or more, scheduled for two or three weekly hemodialysis sessions for a minimum of three months, and having previously undergone hemodialysis for at least six months.

ELIGIBILITY:
Inclusion Criteria:

* Being sixty years or more
* Scheduled for two or three weekly hemodialysis sessions for a minimum of three months
* Having previously undergone hemodialysis for at least six months.

Exclusion Criteria:

* having kidney transplant or peritoneal dialysis, hearing or vision disorders that could impede communication, previous participation in serenity therapy program, and getting psychiatric or psychosocial treatment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Hemodialysis Symptoms Distress-22 scale | 3 months
  The Hemodialysis Symptoms Distress scale-22 (HSD-22) is developed by Chen et al. (2021) to determine the symptom clusters that HD patients experience. It consists of 22 items that are classified into five subscales: sleep disturbance, musculoskeletal discomfort, cardiopulmonary distress, inadequate energy/vitality, and gastrointestinal distress.
Coping Orientation to Problems Experienced Inventory | 3 months
  A 28-item self-report inventory called the Brief COPE Scale was developed by Carver (1997) to assess the various coping mechanisms and responses that an individual may utilize during a stressful life situation including dangerous diseases.
The Emotion Regulation Questionnaire | 3 months
  It is a 10-item questionnaire used to assess participants' tendency to control their emotions using two subscales; cognitive reappraisal (6 items) and expressive suppression (4 items) (Gross& John, 2003).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Hemodialysis unit of the National Medical Institute, Damanhur, El-Behaira Governorate, Egypt.
  - Faculty of Nursing, Alexandria university, Alexandria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abd El Fatah NK, Khedr MA, Elzohairy NW, Harfoush MS, Elgarhy SMA. Effect of serenity therapy on symptoms distress, coping styles, and emotional regulation among geriatric patients undergoing hemodialysis: A randomized controlled trial. Geriatr Nurs. 2026 Jan 21;69:103863. doi: 10.1016/j.gerinurse.2026.103863. Online ahead of print. PMID 41570623